CLINICAL TRIAL: NCT00846417
Title: Impact of ICD Support Groups in Veterans Receiving Internal Cardioverter Defibrillators
Brief Title: Implantable Cardioverter Defibrillator (ICD) Support Groups and Veterans
Status: Terminated | Type: Observational
Why Stopped: No funding, lost support staff, no data collected/processed
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Heather Bloom, Director, Cardiac Electrophysiology Services, Emory University
Other Study IDs: IRB00009530
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2013-09-12 (Estimated); Status verified 2013-09

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia; Sudden Cardiac Death
Keywords: myocardial infarction; heart failure; arrhythmia
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular; Death, Sudden, Cardiac; Myocardial Infarction; Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case: Patients with ICDs who attend the ICD Support Groups.
- Control: Patients with ICDs who do not attend the ICD support groups.

SUMMARY:
In this study, we will compare the quality of life in veterans having ICD who attend the ICD support groups to those who do not. We ask them to answer a set of quality of life questionnaires at baseline and then at 3,6,9 and 12 month visits. These questionnaires would be analyzed to assess if attending support groups made a difference. These results will be compared to a similar study done at Emory University on non veterans.

DETAILED DESCRIPTION:
Sudden cardiac death (SCD) is a major clinical problem, responsible for 400,000 deaths annually in the US(2) Ventricular fibrillation/ventricular tachycardia (VF/VT) is the most common arrhythmia associated with SCD(3). ICD implantation is the only preventive treatment, and clinical trials have clearly established the efficacy of ICD placement for both primary and secondary prevention of SCD(4). Since 1996, ICD implantation has increased dramatically, from 20,000 per year, to 200,000 implanted per year in the US.

Patients are likely to experience varying degrees of psychological, social and physical adjustment both leading up to and following ICD implant. Poor quality of life and depression are common in patients with ICD(5). Anxiety is particularly common, with approximately 24 - 87% of ICD recipients experiencing increased symptoms of anxiety after implantation and diagnostic rates for clinically significant anxiety disorders ranging from 13-38%(6). The occurrence of ICD shocks is generally faulted for this psychological distress, but its causal influence is confounded by the presence of a life threatening medical condition. Depressive symptoms are reported in 24-33% of ICD patients(7). ICD shock related fears are universal and may be the most pervasive psychosocial adjustment challenge ICD patients face.

The literature suggests that ICD recipient QOL is not as high as that among recipients of more benign cardiac devices such as pacemakers. Concerns about ICD shocks and the negative effect of ICDs on patients' sense of control, social interactions, driving, sexuality, capacity to work, and ability to engage in leisure activities appear to adversely influence ICD recipients' perception of health and well being(8).

Support groups are a popular adjunctive treatment for ICD patients because they provide an efficient conduit for patient education spanning the biopsychosocial domains.(9) The active ingredients of support groups probably centre on the universality of many patient concerns and the sharing of information and strategies to deal effectively with these concerns. Dickerson et al found that ICD recipients and their support persons coped with traumatic experience of sudden cardiac death by using story telling in the support group to work through the anxiety and place the event into a manageable explanation(10). Clinical nurse specialist (CNS) - facilitated support group are beneficial if offered, especially if they contact the ICD recipients early during hospitalization and making them aware of this resource(11).

ELIGIBILITY:
Inclusion Criteria:

* Screen for enrollment into 2 groups - ICD support group and non ICD support group, consented, baseline set of QOL questionnaires

Exclusion Criteria:

* Patients that experience varying degrees of psychological, social and physical adjustment both leading up to and following ICD.
* Poor quality of life and depression.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients of primary care cardiology clinics at the Atlanta VAMC
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
All veterans visiting the Atlanta Veterans Administration Medical Center will be screened and enrolled into 2 groups: ICD support group and Non ICD support group. | Documented nine months after the time of enrollment.

SECONDARY OUTCOMES:
This study is observational. It entails questionnaires after enrollment regarding assessing the baseline quality of life in the Veterans on ICDs. | Quality of life questionnaires at 3, 6 and 12 mos follow ups

CONTACTS AND LOCATIONS:
Overall Officials: Heather L Bloom, MD, FACC, Principal Investigator — Emory University IRB